CLINICAL TRIAL: NCT03243890
Title: The Effects of Menaquinone-7 Supplementation in Patients With Aortic Valves Calcification
Brief Title: The Aortic Valve DECalcification (AVADEC) Trial
Acronym: AVADEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Axel Diederichsen (Other)
Responsible Party: Sponsor-Investigator, Axel Diederichsen, Associated professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AVADEC
Record Dates: First submitted 2017-08-02; First posted 2017-08-09 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Aortic Valve Stenosis; Multidetector Computed Tomography; Vitamin K 2; Randomised Clinical Trial
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — menaquinone 7

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 after stratiﬁcation for site, AVC score (300-599 or ≥600) and statin-use. Each site will be provided with sequentially numbered, opaque and sealed envelopes containing randomly generated treatment allocations. Four different types of envelopes are provided; 1) AVC 300-599, no statin-use; 2) AVC 300-599, statin-use; 3) AVC ≥600, no statin-use; and 4) AVC ≥600, statin-use.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization-list is available to the data and safety monitoring board, but patients, nurses, physicians and other data collectors are kept blinded to the allocation during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Study drug. Supplementation with MK-7 (720 µg/day) including the recommended daily dose of vitamin D (25 µg/day)
  Interventions: Dietary Supplement: Menaquinone-7 720 µg/day including the recommended daily dose of vitamin D (25 µg/day).
- Placebo (Placebo Comparator): Placebo tablet (no active treatment). The placebo tablet is matched to the study drug for taste, color, and size.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Menaquinone-7 720 µg/day including the recommended daily dose of vitamin D (25 µg/day). — Half of the patients are randomized to supplementation with MK-7 (720 µg/day) including the recommended daily dose of vitamin D (25 µg/day).
  Arms: Intervention
Dietary Supplement: Placebo — Half of the patients are randomized to placebo treatment (no active treatment).
  Arms: Placebo

SUMMARY:
Aortic stenosis is a common heart valve disease and due to the growing elderly population the prevalence is increasing. The disease is progressive with increasing calcification of the valve cusps. A few attempts with medical preventive treatment have failed, thus presently the only effective treatment of aortic stenosis is surgery. This study will examine the effect of menaquinone-7 (MK-7) supplementation on progression of aortic valve calcification (AVC). The investigators hypothesize that MK-7 supplementation will slow down the calcification process.

ELIGIBILITY:
Inclusion Criteria:

Participants in the Danish Cardiovascular Screening Trial (Trials. 2015 Dec 5;16:554) with an aortic valve calcification score above 300, but without aortic valve stenosis are eligible.

Exclusion Criteria:

* Known aortic valve disease (peak velocity ≥3.0 m/s)
* History of venous thrombosis or other coagulation disorders or use of vitamin K antagonists
* Disorders of calcium and phosphate metabolism
* A life-expectancy < 5 years

Ages: 65 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 389 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Aortic valve calcification | From baseline to two years of follow-up
  The primary endpoint is the change in aortic valve calcification. The natural history of the aortic valve calcification is not adequately understood, and accordingly the changes are analyzed in two prespecified patient subgroups (AVC score 300-599 and ≥600, respectively).

SECONDARY OUTCOMES:
Arterial calcification | From baseline to two years of follow-up
  Change in compiled arterial calcification by non-contrast CT
Aortic size | From baseline to two years of follow-up
  Change in aortic diameter
Coronary plaque composition | From baseline to two years of follow-up
  Change in total plaque burden in the coronaries and carotid arteries by contrast CT
Aortic valve area | From baseline to two years of follow-up
  Change in aortic valve area by transthoracic echocardiography
Bone mineral density | From baseline to two years of follow-up
  Change in bone mineral density as quantitative CT of the columna lumbalis and hip region
Biomarkers of calcification | From baseline to two years of follow-up
  Change in matrix-Gla proteins and osteocalcin with different phosphorylation (p and dp) and carboxylation forms (c and uc).
Quality of life | From baseline to two years of follow-up
  Change in quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Axel CP Diederichsen, PhD, Principal Investigator — Odense University Hospital
Locations (1):
- Department of Cardiology, Odense University Hospital, Odense, Odense C, Denmark

REFERENCES:
- [Background] Lindholt JS, Frandsen NE, Fredgart MH, Ovrehus KA, Dahl JS, Moller JE, Folkestad L, Urbonaviciene G, Becker SW, Lambrechtsen J, Auscher S, Hosbond S, Alan DH, Rasmussen LM, Gerke O, Mickley H, Diederichsen A. Effects of menaquinone-7 supplementation in patients with aortic valve calcification: study protocol for a randomised controlled trial. BMJ Open. 2018 Aug 23;8(8):e022019. doi: 10.1136/bmjopen-2018-022019. PMID 30139903
- [Derived] Diederichsen ACP, Lindholt JS, Moller S, Ovrehus KA, Auscher S, Lambrechtsen J, Hosbond SE, Alan DH, Urbonaviciene G, Becker SW, Fredgart MH, Hasific S, Folkestad L, Gerke O, Rasmussen LM, Moller JE, Mickley H, Dahl JS. Vitamin K2 and D in Patients With Aortic Valve Calcification: A Randomized Double-Blinded Clinical Trial. Circulation. 2022 May 3;145(18):1387-1397. doi: 10.1161/CIRCULATIONAHA.121.057008. Epub 2022 Apr 25. PMID 35465686
- See also: Protocol — https://bmjopen.bmj.com/content/8/8/e022019.long

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-24): https://cdn.clinicaltrials.gov/large-docs/90/NCT03243890/SAP_000.pdf